CLINICAL TRIAL: NCT00888901
Title: Assessment of Platelet Function in Patients With Chronic Autoimmune Thrombocytopenic Purpura (cAITP) Treated With the Thrombopoietin Receptor (MPL) Agonist Eltrombopag.
Brief Title: Platelet Function in Idiopathic Thrombocytopenic Purpura (ITP) Patients With Eltrombopag
Acronym: PLATEFUN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ingrid Pabinger, MD (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Ingrid Pabinger, MD, Univ.-Prof. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IP-001; Eltrombopag 112650
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: ITP; eltrombopag; platelet function; thrombocytopenia; Platelet function in patients with cAITP on eltrombopag
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — eltrombopag; Adrenal Cortex Hormones; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Patients on eltrombopag
  Interventions: Drug: eltrombopag
- 2 (Active Comparator): Patients on corticosteroids
  Interventions: Drug: corticosteroids (Aprednislon)
- 3 (No Intervention): Untreated patients

INTERVENTIONS:
Drug: eltrombopag — eltrombopag tablets daily, in increasing dosage, for three months
  Other Names: SB-497115-GR, Promacta (USA), Revolade (EU)
  Arms: 1
Drug: corticosteroids (Aprednislon) — corticosteroids in decreasing dosage
  Other Names: Aprednislon
  Arms: 2

SUMMARY:
This is a single-center, prospective, controlled study with one eltrombopag treatment group and 2 control groups, one on standard steroid treatment, and another one untreated.

The aim of the study is to determine the effect of Thrombopoietin Receptor (MPL) agonists on shear-induced platelet activation.

DETAILED DESCRIPTION:
STUDY DESIGN:

Single-center (Medical University Vienna), prospective, controlled study. Patients will be recruited at the Division of Haematology and Haemostaseology at the Medical University in Vienna, one eltrombopag treatment group and 2 control groups, one on standard steroid treatment, another one untreated.

AIM OF THE STUDY:

To determine the effect of MPL agonists on shear-induced platelet activation. Data obtained from patients treated with eltrombopag shall be compared to those from untreated patients and patients on steroids. These investigations will extend previous studies that investigated platelet function without in vitro activation in patients receiving eltrombopag.

PATIENTS:

Trial Population:

Total number of patients n=34: 12 on eltrombopag, 12 on corticosteroids and 10 without treatment will be included in this trial.

Treatment with eltrombopag or corticosteroids. Eltrombopag starting dose: 25 mg/day, increased as needed (to 50 mg or maximum 75 mg once daily) every 2 weeks to reach a platelet count between 50,000-100000/µL and tapering the dosis if platelet count >= 100,000/µL. Afterwards, if platelet count stable (tolerance +/- 20%), platelet control every 4 weeks, otherwise weekly.

Prednisolone starting dose: 1 mg/kg/day to reach a platelet count between 50,000-100,000 /µL tapering of the dosage if platelet count >= 100,000/µL.

Laboratory Investigations:

In the eltrombopag group and in the newly treated prednisolone group platelet counts and platelet function tests will be performed at planned visits.

In patients who are on continuous corticosteroids (part of control group I) and untreated patients (control group II), which have a platelet count between 50,000 and 100,000/µL platelet counts, reticulated platelets, platelet function tests and platelet antibodies will be studied at entry and after 4 weeks (+ 5 days).

ELIGIBILITY:
Inclusion Criteria (for all groups):

* Male and female patients with an established chronic autoimmune thrombocytopenia (cAITP)
* Age ≥ 18 and ≤ 90 years
* Females, if not pregnant, not nursing and consenting to perform safe anti-contraception
* Written consent before any study related procedure

Inclusion Criteria (for patients treated with eltrombopag):

* Platelet count < 50,000 /µL at screening
* At least one prior alternative cITP therapy

Inclusion Criteria (for patients treated with corticosteroids - Control group 1):

* Platelet count < 50,000 /µL in history
* At least 50% of the patients should have < 50,000 /µL at inclusion and should be followed for 3 months

Inclusion Criteria (for patients untreated - Control group 2):

* Platelet count < 50,000 /µL in history
* At screening platelet count between 50,000 and 100,000 /µL

Exclusion Criteria (for all patients):

* History of venous or arterial thromboembolism or stroke
* Known coronary heart disease or cardiac arrythmias
* Known HIV or Hepatitis C infection
* Impaired liver function defined as elevated ALT > 1.5 UNL, bilirubin more than ULN, albumin less than normal value
* Prothrombin time less than normal value
* Elevated creatinine level (> 1.3 ULN)
* Unable/unwilling to follow protocol
* Previous or active malignancy
* Patients who have been included in any other study with eltrombopag any time before
* Patients treated with another investigational product within the last 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The shear-induced platelet activation (SC) is considered as the primary outcome measure. | After an average of 2-4 weeks, when patient has a platelet count between 50,000 and 100,000/µL.

SECONDARY OUTCOMES:
Rise of reticulated platelets and variation of platelet antibodies. | After an average of 2-4 weeks, when patient has a platelet count between 50,000 and 100,000/µL.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Pabinger, Prof. Dr., Principal Investigator — Medical University of Vienna

REFERENCES:
- [Derived] Haselboeck J, Kaider A, Pabinger I, Panzer S. Function of eltrombopag-induced platelets compared to platelets from control patients with immune thrombocytopenia. Thromb Haemost. 2013 Apr;109(4):676-83. doi: 10.1160/TH12-07-0522. Epub 2013 Feb 7. PMID 23389750
- See also: Division of hematology and hemostaseology, Med. Univ. Vienna — http://www.meduniwien.ac.at/haematology/